Efficacy of the Transition of the Foot Strike Pattern From Rearfoot to Midfoot or Forefoot During Running on Pain and Disability in Cadets With Chronic Musculoskeletal Pain

NCT ID not yet assingned

## **Statistical Analysis Plan**

The analysis of the information will be conducted by a researcher who will provide coded data, and an entire analysis will be performed by the principle of intention of treatment. A description is appropriate to present as the characteristic of the participants in the three groups. The Shapiro-Wilk test and the numerical variables with the normal distribution of data through media and standard deviations or through mediations and interquartile ranges will be performed when there is no normal distribution. Variables can be separated by proportions and number of participants. The trend effect analysis was performed using mixed linear models. The analysis of unrealized time-averaging potential was performed using causal mediation methods, with a 95% confidence interval (95% CI). All analyzes are based on Rstudio version 3.5.0 (Foundation for Computational Statistics, Vienna, Austria